CLINICAL TRIAL: NCT02150369
Title: Investigating Cognitive/Affective/Sleep Symptoms During High-dose Interleukin-2 Therapy
Brief Title: Interleukin-2-Induced Cognitive/Affective/Sleep Symptoms
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00053989
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Renal Cell Carcinoma; Metastatic Melanoma; High-dose Interleukin-2
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient, care partner, primary nurse case: In Phase I of this pilot, a case is comprised of the metastatic RCC patient receiving IL-2, their care partner, and their primary nurse. In Phase II, the IL-2 patient can either have MM or metastatic RCC. The care partner for this study will be the family member or friend staying with the IL-2 patient throughout treatment.

SUMMARY:
-Purpose: Phase I: To test the methods, data collection and analysis in a study to evaluate cognitive/affective/sleep symptoms in one patient undergoing treatment with high-dose Interleukin-2 (IL-2) for metastatic renal cell carcinoma (RCC), their informal caregiver and their primary nurse.

Phase II: A pilot study examining up to 10 IL-2 cases to describe cognitive/affective/sleep symptoms of patients receiving high-dose IL-2 therapy for metastatic melanoma (MM) or metastatic RCC in order to develop interventional studies to minimize these symptoms.

-Aims: In this pilot, a case is comprised of the metastatic RCC patient receiving IL-2, their care partner, and their primary nurse. The care partner for this study will be the family member or friend staying with the IL-2 patient throughout treatment.

Phase I (Evaluation of Methods and Procedures):

One case will be examined to evaluate the methods, data collection and analysis to be used in this study. The aims of Phase I of this study are to: Aim 1) Evaluate recruitment and enrollment procedures to enroll one IL-2 case, comprised of the IL-2 patient, their care partner and their primary nurse; Aim 2) Evaluate administration procedures, data collected, and analysis of four questionnaire scales to detect the trajectory of cognition [Attentional Function Index and Montreal Cognitive Assessment] and affect [Hamilton Anxiety scale and Inventory of Depressive Symptomatology-Clinician] in the IL-2 patient from the start to the end of a cycle of treatment; Aim 3) Evaluate procedures, data collected and analysis of journal entries from the care partner who are to record their thoughts, observations, and feelings concerning any changes in the patient's behavior or cognition during IL-2 treatment every 8 hours; Aim 4) Evaluate procedures, data collected and analysis of semi-structured questionnaires completed by the primary nurse taking care of the patient receiving IL-2 which will describe any changes in behavior or cognition in the patient during their IL-2 treatment; and Aim 5) Evaluate procedures, data collected and analysis of data of interviews with the IL-2 patient to further discern what symptoms endorsed on the measurement scales represent and how they are characterized, and interviewing the primary nurse to gain any additional data on cognitive/affective symptoms observed in the IL-2 patient.

Phase II (Investigating Cognitive, Affective and Sleep Alterations in Patients Receiving high dose IL-2 therapy): Up to 10 additional cases will be enrolled to understand cognitive, affective and sleep symptoms induced from IL-2 therapy in oncology patients with MM or metastatic RCC, and help design future studies to ameliorate these treatment-limiting symptoms. The specific aims of this study are to: Aim 1) Describe cognitive (language, concentration, mental fatigue, confusion, attention, short-term memory, and orientation), affective (depression, anxiety, mood alterations), and sleep disturbance symptoms in patients receiving 1 to 4 cycles (up to 8-weeks) of high-dose IL-2 therapy. Aim 2) Examine observed patient experiences of cognitive/affective/sleep symptoms from each patient's primary care partner, and primary nurse during 1 to 4 cycles of IL-2 therapy. Aim 3) Describe the trajectories of cognitive/affective/sleep symptoms in patients with MM or metastatic RCC undergoing 1 to 4 cycles of IL-2 therapy. Not all patients will receive 4 cycles of IL-2, because treatment will depend on a) disease progression and b) side effect toxicity; therefore, the symptom trajectory will be described for the cycles completed in situations where all cycles are not completed.

DETAILED DESCRIPTION:
-Background & Significance: Alterations in cognitive, affective and sleep functioning are among the most challenging side effects experienced by 80% of patients undergoing high dose IL-2 therapy. Altered cognition includes a wide array of symptoms such as changes in concentration, attention, short-term memory, confusion, mental fatigue, executive functioning, abstraction, language, basic arithmetic, and orientation. Affective symptoms include mood alterations, depression, anxiety, psychosis, hallucinations, aggression, suicidal ideation, and coma. Sleep symptoms include the insomnias (initial, middle, delayed) and hypersomnia. Severe cognitive/affective/sleep symptoms may result in early termination of IL-2 therapy, preventing the patient from receiving its full benefits. In some patients, cognitive, affective and sleep symptoms continue throughout the remainder of their life, decreasing the quality of life for patients and their families. Although prior investigators reported chemotherapy-related altered cortical and cognitive function including slowed processing time and decreased brain activation, as well as signs of increased cytokines and decreased gray matter, studies investigating the trajectory of immunotherapy-related altered cognition have not been found in published literature. Describing the impact of IL-2 therapy on cognition, affect and sleep is essential to designing interventions to ameliorate these treatment-limiting symptoms. Because IL-2 patients receive several doses of medication over a number of days, exploring these symptoms through a trajectory analysis of these symptoms is critical. Without fully understanding the breadth and depth of IL-2-induced cognitive/affective/sleep symptoms, advances in science to alleviate these symptoms are at a standstill.

Metastatic RCC and MM are two cancers treated with IL-2, where surgery, chemotherapy and radiation therapy are ineffective for patients with stage III and IV disease. For phase I of this pilot study, we will focus only on enrolling one IL-2 patient with metastatic RCC, their care partner and their primary nurse; as many five subjects comprising one case may be recruited for consent. In 2014, the National Cancer Institute estimates 76,000 new diagnoses and 9,700 deaths secondary to melanoma, and 64,000 new cases and 14,000 deaths secondary to kidney cancer. IL-2, a cytokine based immunotherapy, is administered to patients with metastatic disease to stimulate their immune systems to fight off cancerous cells, and is one of the few treatments available for patients with progressed disease. When IL-2 is administered in high-dose, intravenous form, patients experience severe and potentially life-threatening side effects. The long-term impact of IL-2 treatments on cognitive/affective symptoms has not been documented. Despite severe symptoms and side effects, 33% of MM patients have some response to IL-2 treatment and 15% of MM patients show a complete response with no detectable metastases after treatment. In RCC, 14% of patients show some response and 8% show a complete response. Thus, interventions that help patients complete treatment are warranted and would build on knowledge gained in this study.

-Procedures: Phase I will enroll a case over one cycle of high-dose IL-2 given over five days. Phase II will enroll up to 10 additional cases for up to four cycles of high-dose IL-2 therapy. High-dose IL-2 is defined as 600,000-720,000 International Units/kilogram, administered intravenously over 15 minutes, every 8 hours for a maximum of 14 consecutive doses; these 14 doses comprise one treatment cycle. Quantitative data will be collected using questionnaires administered to the IL-2 patient measuring cognitive/affective/sleep symptoms before and after each cycle of high-dose IL-2 to describe any longitudinal changes in the patient over the therapy course. Qualitative data will be collected through semi-structured journal entries written by the care partner, semi-structured questionnaires given to the nurses after each dose of IL-2, and interviews with the IL-2 patient, care partner and primary nurse.

Three constructs (cognitive symptoms, affective symptoms, sleep symptoms) will be used to describe IL-2-induced cognitive/affective/sleep symptoms using four sources for data collection (the IL-2 patient, their primary care partner, their nurses, and their primary nurse). The index participant will receive up to three high-dose IL-2 treatments per day, at 8-hour intervals, for a maximum of 14 doses per cycle. The pattern of data collection in Phase I will repeat for a maximum of four IL-2 cycles in Phase II.

Cognitive/affective/sleep symptoms experienced by the patient will be evaluated using six scales. Scales will be administered to the index participant upon their admission to the hospital before receiving the first dose of IL-2 in each cycle, and 16-hrs after the last IL-2 dose for each cycle. The nurse caring for the IL-2 patient will be contacted over the phone and we will be in constant communication about the timing of IL-2 administration and therapy ending. Questionnaires will be administered in the patient's private hospital room. Although it would be ideal to administer these surveys following each IL-2 dose, the IL-2 patient is disrupted every four hours for IL-2 related care. Administering the scales only twice during each cycle will reduce patient burden and will be sufficient to assess for longitudinal changes in cognitive/affective/sleep symptoms. For symptoms endorsed by the patient 16-hr post-treatment, we will interview the IL-2 patient to further discern what these symptoms represent and how they are characterized. This semi-structured interview will be recorded and transcribed.

The care partner will be asked to record observations of the patient's cognitive, affective and sleep symptoms as a journal entry three times per day, prior to the first IL-2 dose and then after each dose. The semi-structured journal entry will contain a checklist to signify when symptoms are observed by the care partner, such as the patient pulling out catheters or intravenous lines, confusion, hallucinating, signs of depression, and/or anxiety. The checklist will be followed by a prompt that will read, "For the boxes you checked above, please describe the changes you witnessed. When did the symptom appear? How long did the symptom last? How severe is the symptom? Can you describe the situation? Did anything make this symptom better or worse?" Following this prompt, the final open-ended prompt will read, "If there are other changes in the patient that you feel the team should know about, please feel free to write about these changes as well." After treatment has ended, the care partner will participate in a post-treatment semi-structured interview at the end of each cycle of therapy. This interview will be recorded and transcribed.

Similar to the care partner, nurses that participate in the patient's care will receive the same semi-structured prompt as the care partner. Nurses will also be asked to write, 'I did not witness any cognitive or affective changes in the IL-2 patient during my time with the patient' if changes in symptoms were not observed. A folder containing the prompt for the nurses will be kept in a secure place on the unit for the nurses to access so they can retrieve a form containing the prompt prior to doing their nursing assessment. The nurses will be encouraged to complete the form after each IL-2 infusion. Once the primary nurse for the IL-2 patient is identified, we will approach s/he for consent and interview the primary nurse to gain any additional data on cognitive/affective/sleep symptoms observed in the IL-2 patient. This interview will be recorded and transcribed. Field notes will be collected throughout the study to enrich the data. Collection of data from multiple sources such as interviews, journal entries and field notes will allow for a comprehensive understanding of the data.

ELIGIBILITY:
Inclusion Criteria (of the IL-2 patient):

* Persons diagnosed with metastatic RCC/MM (stage III or stage IV) disease
* 18-65 years of age
* English speaking and literate
* Receiving HD IL-2 (720,000 IU/kg of IL-2 IV q8hr for a total of 14 doses per cycle) therapy at Duke University Hospital
* Must have a care partner (family member or friend) active in their care during IL-2 treatments

Exclusion Criteria:

* Previously documented cognitive disorder
* Congenital brain defects
* Traumatic brain injuries

Primary care partner: defined as the primary family member or friend who will be staying with the patient at the hospital during the patient's IL-2 therapy OR is active in the patient's care. The IL-2 patient may have up to two primary care partners, for example a care partner for nights/days or alternating days. Care partners who are under 18 years may enroll if their parent is the IL-2 patient. For this study, the care partner must be at least 16 years old in order to participate because of the nature of the study. Their parent must be present and must consent for enrollment.

Primary Nurse: will be identified by the unit or self-identified as the nurse who best "knows" the patient and his/her care. The primary nurse must be a Registered Nurse.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants will be recruited from Duke University Hospital (Duke North) in Durham, NC.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Participant enrollment | 6 months
  Phase I: Participant enrollment will be evaluated by determining the difficulty of recruitment and enrollment of one case, comprised of the IL-2 patient, their care partner and their primary nurse. To determine enrollment difficulty, the time taken to enroll one case will be recorded.

SECONDARY OUTCOMES:
Participant burnout | 1 months
  Phase I: The IL-2 patient, their care partner and their primary nurse will be evaluated for participant burnout. This will be assessed by evaluating participant retention throughout the duration of the study. We will look at if the IL-2 participant, their care partner, and their primary nurse stayed enrolled for the duration of the study.

OTHER OUTCOMES:
Participant burden | 1 months
  Phase I: The IL-2 participant will be evaluated to determine if all four scales (HAM-A, AFI, IDS, MoCA) were completed at the start and end of each IL-2 cycle. The time required to complete these four scales will be recorded to determine patient burden.
  The care partner will be evaluated based on how many of the written journal entries they were able to complete. Journal entries are written at the start of treatment, and every eight hours throughout treatment (maximum of 15 entries). The time required to complete these written entries will also be evaluated.
  Finally, nurse(s) will be evaluated based on whether they were able to respond to the short-response, open-ended question during their work day, while the primary nurse will be evaluated in their willingness to participate in a recorded interview at the end of the treatment cycle.
Cognitive Symptoms I | 4 months
  Phase II: Cognitive symptoms will be measured by quantitative scores on the Montreal Cognitive Assessment completed by the patient receiving IL-2 during hospitalization.
Cognitive Symptoms II | 4 months
  Phase II: Cognitive symptoms will be measured by quantitative scores on the Attentional Function Index completed by the patient receiving IL-2 during hospitalization.
Cognitive Symptoms III | 4 months
  Phase II: Cognitive symptoms will be measured by qualitative reports of symptom change through journal entries written by the care partner during hospitalization.
Cognitive Symptoms IV | 4 months
  Phase II: Cognitive symptoms will be measured by qualitative reports of symptom change through interviews during hospitalization.
Affective Symptoms I | 4 months
  Phase II: Affective symptoms will be measured by quantitative scores on the Inventory of Depressive Symptomatology-Clinican completed by the patient receiving IL-2 during hospitalization.
Affective Symptoms II | 4 months
  Phase II: Affective symptoms will be measured by quantitative scores on the Hamilton Anxiety Scale completed by the patient receiving IL-2 during hospitalization.
Affective Symptoms III | 4 months
  Phase II: Affective symptoms will be measured by qualitative reports of symptom change through journal entries written by the care partner during hospitalization.
Affective Symptoms IV | 4 months
  Phase II: Affective symptoms will be measured by qualitative reports of symptom change through interviews during hospitalization.
Sleep Symptoms I | 4 months
  Phase II: Sleep symptoms will be measured by quantitative scores on the Inventory of Depressive Symptomatology-Clinican completed by the patient receiving IL-2 during hospitalization.
Sleep Symptoms II | 4 months
  Phase II: Sleep symptoms will be measured by qualitative reports of symptom change through journal entries written by the care partner during hospitalization.
Sleep Symptoms III | 4 months
  Phase II: Sleep symptoms will be measured by qualitative reports of symptom change through interviews during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Robin B. Knobel, PhD, RN, Principal Investigator — Duke University; Donald E. Bailey, PhD, RN, FAAN, Study Chair — Duke University; Tara K. Mann, RN, Study Chair — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

REFERENCES:
- See also: RCC and high-dose IL-2 — http://www.cancernetwork.com/renal-cell-carcinoma/high-dose-interleukin-2-therapy-metastatic-renal-cell-carcinoma-and-metastatic-melanoma-still